CLINICAL TRIAL: NCT00145405
Title: Comparable Effects of Lanreotide Autogel and Octreotide LAR on GH, IGF-I Levels and Patient Satisfaction - A Twelve Month Randomized Cross-Over Study in Patients With Acromegaly
Brief Title: Comparable Effects of Lanreotide Autogel and Octreotide LAR on GH, IGF-I Levels and Patient Satisfaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 009
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Acromegaly
Keywords: Acromegaly; somatostatin analogues; lanreotide; octreotide; GH; IGF-I; injection site
MeSH Terms: conditions — Acromegaly

INTERVENTIONS:
Drug: Lanreotide Autogel and Octreotide LAR

SUMMARY:
The morbidity and the mortality in acromegalic patients closely correspond to growth hormone (GH) levels and therefore efficient long-term treatment is important.

Neurosurgery is the first choice of treatment in acromegalic patients. Surgery normalizes GH levels in about 80% of patients with microadenomas, but less than 50 % of patients with macroadenomas respond sufficiently to surgery alone. In most patients, additional medical therapy is therefore needed.

Somatostatin analogues have successfully been used in treatment of acromegaly if surgery or radiotherapy can not lead to normal GH and IGF-I levels. Lanreotide Autogel (LAN) is a new formulation of lanreotide consisting of a prolonged release aqueous formulation, which can be injected intramuscularly or deep subcutaneously once every 28 days.

Aim

The aim of the present study was to compare the efficacy of OCT and LAN in obtaining GH and IGF-I levels according to the 2000 Consensus. Furthermore, we wanted to evaluate which treatment modality resulted in the lowest possible IGF-I and GH levels and the highest patient satisfaction.

DETAILED DESCRIPTION:
Introduction The morbidity and the mortality in acromegalic patients closely correspond to growth hormone (GH) levels and therefore efficient long-term treatment is important (1).

Neurosurgery is the first choice of treatment in acromegalic patients. Surgery normalizes GH levels in about 80% of patients with microadenomas, but less than 50 % of patients with macroadenomas respond sufficiently to surgery alone (1). In most patients, additional medical therapy is therefore needed.

Somatostatin analogues have successfully been used in treatment of acromegaly if surgery or radiotherapy can not lead to normal GH and IGF-I levels (2, 3, 4, 5). Lanreotide Autogel (LAN) is a new formulation of lanreotide consisting of a prolonged release aqueous formulation, which can be injected intramuscularly or deep subcutaneously once every 28 days.

Aim The aim of the present study was to compare the efficacy of OCT and LAN in obtaining GH and IGF-I levels according to the 2000 Consensus. Furthermore, we wanted to evaluate which treatment modality resulted in the lowest possible IGF-I and GH levels and the highest patient satisfaction.

Inclusion criteria

* all the patients which receive octreotide LAR can be included;
* new diagnosed patients with clinical and biochemical acromegaly , if medicine therapy is indicated;
* as long as they do not fit in the exclusion criteria. Exclusion criteria
* which had not given their consent after they received standard information about the study;
* current malign disease;
* somatostatin analogues intolerance;
* elevation of lever enzymes;
* pregnancy.

Design The study is designed as a randomized cross-over trial. Patients will be randomized to receive either OCT or LAN for 6 months and will be then changed to the opposite therapy for 6 months without interruption between the two therapies Both OCT and LAN will be administered once every 28 days. OCT will be given intramuscularly and LAN deep subcutaneously by the patients' general practitioner or by a study nurse. At times 0, 4, 6, 10, and 12 months, the patients will be attended for clinical evaluation, at the department of Endocrinology, Odense University Hospital.

Patients previously treated with OCT will receive unchanged doses of OCT during the study period and OCT dose will use to calculate LAN doses. The administered OCT dose will be determined as the dose necessary to obtain normal IGF-I levels and/or GH<1mU/l (<0.4 μg/ l) or alternatively the highest tolerated dose.

The LAN doses will be calculated using the OCT doses as follows: 10 mg OCT ≈ 60 mg LAN; 20 mg OCT ≈ 90 mg LAN; 30 mg OCT ≈ 120 mg LAN.

Evaluation program (at 0, 4, 6, 10, 12 months) Clinical evaluation: weight, blood pressure, inspection of the injection site and evaluation of possible side effects.

Analyses: GH and IGF-I, prolactin, thyroid hormone, oestrogen, testosterone, LH, and FSH, fasting plasma glucose and glycosylated hemoglobin, liver enzymes levels.

The study will be supported by Beaufor Ipsen Industry and further technical assistance will be supplied by Endocrinology Department, Odense University Hospital.

References

1. Giustina, A., Barkan, A., Casanueva, F. F., Cavagnini, F., Frohman, L., Ho, K., Veldhuis, J., Wass, J., Von, Werder K., and Melmed, S. Criteria for cure of acromegaly: a consensus statement.J.Clin.Endocrinol.Metab 2000 85 526-529
2. Chanson, P. Somatostatin analogs in the treatment of acromegaly: the choice is now possible.Eur.J.Endocrinol. 2000 143 573-575
3. Cozzi, R., Dallabonzana, D., Attanasio, R., Barausse, M., and Oppizzi, G. A comparison between octreotide-LAR and lanreotide-SR in the chronic treatment of acromegaly.Eur.J.Endocrinol. 1999 141 267-271
4. Turner, H. E., Vadivale, A., Keenan, J., and Wass, J. A. A comparison of lanreotide and octreotide LAR for treatment of acromegaly.Clin.Endocrinol.(Oxf) 1999 51 275-280
5. Verhelst, J. A., Pedroncelli, A. M., Abs, R., Montini, M., Vandeweghe, M. V., Albani, G., Maiter, D., Pagani, M. D., Legros, J. J., Gianola, D., Bex, M., Poppe, K., Mockel, J., and Pagani, G. Slow-release lanreotide in the treatment of acromegaly: a study in 66 patients.Eur.J.Endocrinol. 2000 143 577-584

ELIGIBILITY:
Inclusion Criteria:

* All the patients which receive octreotide LAR can be included;
* New diagnosed patients with clinical and biochemical acromegaly , if medicine therapy is indicated;
* As long as they do not fit in the exclusion criteria.

Exclusion Criteria:

* Which had not given their consent after they received standard information about the study;
* Current malign disease;
* Somatostatin analogues intolerance;
* Elevation of lever enzymes;
* Pregnancy.

Ages: 22 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2002-09; Study Completion 2004-12

PRIMARY OUTCOMES:
GH and IGF-I levels after 4, 6, 10, 12 months therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark